CLINICAL TRIAL: NCT01317784
Title: Behavioral Science Aspects of Rapid Test Acceptance
Acronym: BSARTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, Long Beach (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Dennis G. Fisher, Professor and Director, California State University, Long Beach
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 07373710; R01DA030234 (NIH)
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: HIV; Hepatitis C; Hepatitis B; Syphilis
Keywords: diagnosis screening; HIV serodiagnosis; HCV antibodies; serologic tests; Bedside testing; diagnostic test kits; syphilis serodiagnosis
MeSH Terms: conditions — Hepatitis C; Hepatitis B; Syphilis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- All tests. (Experimental): Choose from all 16 possible tests.
  Interventions: Device: Rapid tests for HIV, HCV, HBV, and syphilis
- HIV/HCV (Active Comparator): Choice of 10 different HIV and hepatitis C tests in the bundle.
  Interventions: Device: HIV/HCV
- HIV/Syphilis (Active Comparator): Choice of 7 different tests for HIV and syphilis.
  Interventions: Device: HIV/syphilis
- HIV only (Active Comparator): Choice of 4 rapid tests for HIV only.
  Interventions: Device: HIV only

INTERVENTIONS:
Device: Rapid tests for HIV, HCV, HBV, and syphilis — Choice of 16 different rapid tests. Only 12 manufacturer and names are shown because some are used with both blood and oral fluid. When they are used on both specimens, they are counted as two tests.
  Other Names: INSTITM HIV-1 Antibody Test (bioLytical Laboratories, Inc.); Determine HIV-1/2 Ag/Ab Combo (Alere, Inc.); DPP® HIV 1/2 Screen Assay (Chembio, Inc.); OraQuick HCV antibody test (Orasure); DPP® HCV Screen Assay (Chembio, Inc.); DPP® HIV-HCV Screen Assay (Chembio, Inc.); Multiplo Rapid HIV/HCV Antibody Test (MedMira, Inc.); DPP® Syphilis Screen & Confirm Assay (Chembio, Inc.); DPP® HIV-Syphilis Screen Assay (Chembio, Inc.); DPP® HIV-HCV-Syphilis Screen Assay (Chembio, Inc.); Multiplo Rapid HIV/HCV/HBV Antibody Test (MedMira, Inc.)
  Arms: All tests.
Device: HIV/HCV — Choice of 10 different tests for HIV and hepatitis C.
  Other Names: INSTITM HIV-1 Antibody Test (bioLytical Laboratories, Inc.); Determine HIV-1/2 Ag/Ab Combo (Alere, Inc.); DPP® HIV 1/2 Screen Assay (Chembio, Inc.); OraQuick HCV antibody test (Orasure); DPP® HCV Screen Assay (Chembio, Inc.); DPP® HIV-HCV Screen Assay (Chembio, Inc.); Multiplo Rapid HIV/HCV Antibody Test (MedMira, Inc.)
  Arms: HIV/HCV
Device: HIV/syphilis — Choice of 7 different tests for HIV and syphilis
  Other Names: INSTITM HIV-1 Antibody Test (bioLytical Laboratories, Inc.); Determine HIV-1/2 Ag/Ab Combo (Alere, Inc.); DPP® HIV 1/2 Screen Assay (Chembio, Inc.); DPP® Syphilis Screen & Confirm Assay (Chembio, Inc.); DPP® HIV-Syphilis Screen Assay (Chembio, Inc.)
  Arms: HIV/Syphilis
Device: HIV only — Choice of 4 different tests for HIV only.
  Other Names: INSTITM HIV-1 Antibody Test (bioLytical Laboratories, Inc.); Determine HIV-1/2 Ag/Ab Combo (Alere, Inc.); DPP® HIV 1/2 Screen Assay (Chembio, Inc.)
  Arms: HIV only

SUMMARY:
The relevance of this research to public health is to make it possible to test for hepatitis C and syphilis at point of care so that people will receive their results immediately instead of requiring people to wait for at least a week to get their test results. This research will make rapid tests for HIV available that can detect HIV infection earlier and are more accurate than current tests available in the United States.

DETAILED DESCRIPTION:
This application addresses "Studies to improve access and utilization of HIV counseling and testing" for "HIV/AIDS and AIDS-related co-infections" such as "hepatitis C virus (HCV), other sexually transmitted infections (STIs)" that are part of PA-07-307 Drug Abuse Aspects of HIV/AIDS. The only rapid tests that are approved for use in the US currently are for HIV infection. Tests for other conditions such as hepatitis C (HCV) and syphilis are in use in other countries. In response to an Opportunity that the CDC published in the Federal Register, there are now candidate rapid test kits for HCV and syphilis available for experimental use in the US. Different combinations of rapid and standard tests will be offered to participants in a four-arm trial to assess which tests are accepted by the participants. Only a minority of clients at CBRS who have been offered the rapid test for HIV have accepted it. Those who chose rapid HIV tests were more likely to be male, educated, gay, young and White. They were less likely to be Black, or injection drug users. The proposed study has the potential to have a significant impact upon screening for HIV, syphilis, and HCV. Rapid tests have the potential to increase the receipt of test results, particularly among groups that are less likely to return for their results using traditional testing. The candidate tests are designed for Point of Care (either oral fluid and/or whole blood), and thus will require real-time testing, so the trial will be able to evaluate both the accuracy of the tests in settings of intended use and their acceptability to potential clients in real-world situations.

ELIGIBILITY:
Inclusion Criteria:

* Over 17 years old
* Mentally stable
* Sober
* Able to understand English or Spanish
* At least one good vein for phlebotomy
* Member of Behavioral Risk Group

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2011-05; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Test choice profile | one day (day one of study)
  Which tests do participants choose to receive when bundled in different combinations?

SECONDARY OUTCOMES:
Return for standard test results | one week
  Is there a different return for test results rate for the different arms of the study?

CONTACTS AND LOCATIONS:
Overall Officials: Dennis G Fisher, Ph.D., Principal Investigator — California State University, Long Beach
Locations (1):
- Center for Behavioral Research and Services, Long Beach, California, United States